CLINICAL TRIAL: NCT03906097
Title: The Effects of Play and Competition-Based Cognitive Therapy on Executive Functions and Occupational Routines in Children With Dyslexia
Brief Title: The Effects of Play and Competition-Based Cognitive Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Gokcen Akyurek, PhD PT, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-375
Record Dates: First submitted 2019-04-04; First posted 2019-04-08 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Dyslexia; Executive Dysfunction
Keywords: Dyslexia; Executive function; Cognitive control; Inhibition; Working memory; Prefrontal Cortex
MeSH Terms: conditions — Dyslexia; Inhibition, Psychological

STUDY DESIGN:
Intervention Model Description: Before randomization, 80 children were performed the tests (TVPS-3 and DOTCA-Ch) and questionnaires (BRIEF and EFORTS) were given to their parents and teachers. Then, SPSS 24.00 was randomized with the program and the control group was divided into 2 equal groups (intervention group n = 40; control group n = 40). The intervention group was received cognitive therapy for 10 weeks, 3 days a week, 1 hour per day; the control group was the group who continued the special education program (Figure 3.1). Both groups were evaluated three times at baseline, at the end of the 10th week and at the end of the third month (follow up).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): SPSS 24.00 was randomized with the program and the control group was divided into 2 equal groups (intervention group n = 40; control group n = 40). The intervention group was received cognitive therapy for 10 weeks, 3 days a week, 1 hour per day; the control group was the group who continued the special education program (Figure 3.1). Both groups were evaluated three times at baseline, at the end of the 10th week and at the end of the third month (follow up).
  Interventions: Other: Play and Competition-Based Cognitive Therapy
- control (No Intervention): SPSS 24.00 was randomized with the program and the control group was divided into 2 equal groups (intervention group n = 40; control group n = 40). The intervention group was received cognitive therapy for 10 weeks, 3 days a week, 1 hour per day; the control group was the group who continued the special education program (Figure 3.1). Both groups were evaluated three times at baseline, at the end of the 10th week and at the end of the third month (follow up).

INTERVENTIONS:
Other: Play and Competition-Based Cognitive Therapy — The intervention group was received play and competition-based cognitive therapy for 10 weeks, 3 days a week, 1 hour per day; the control group was the group who continued the special education program
  Arms: intervention

SUMMARY:
Purpose: The aim of this study was to investigate the effects of play and competition-based cognitive therapy (PCB-CT) on executive function and occupational routines in children with dyslexia.

Method: In this randomized control trail, 64 children with dyslexia (between 7-12 ages) were randomly selected from the 162 clients who applied to the clinic. Children were divided randomly into a treatment group and a control group. Children in the intervention group was given cognitive therapy for 10 weeks, 3 days a week for one hour sessions while no therapy was received to the control group. In order to evaluate the cognition of the children Test of Visual Perceptual Skills-3 (TVPS-3) and Dynamic Occupational Therapy Cognitive Assessment (DOTCA-Ch), to evaluate executive functions the Behavior Rating Inventory of Executive Function (BRIEF) and to evaluate occupational routine The Executive Functions and Occupational Routines Scale (EFORTS) were used. The evaluations were done at baseline, after treatment and the end of the 3rd month for both groups.

DETAILED DESCRIPTION:
The participants included in this study if they had only dyslexia diagnosis, aged between 7-12 years and had a 90 and above IQ score (normal IQ), in addition didn't have multiple conditions (neurological problems such as epilepsy) or primary psychiatric comorbidities (i.e. depression, anxiety, psychosis).

Test of Visual Perceptual Scale-3(TVPS-3); The TVPS-3 was originally designed for children but the author Dr. Gardner also reported statistically significant differences between three groups diagnosed as having either developmental delay, head injury or learning disability. This test in its third edition has been revised by Martin for appropriate use in an adult population, with scores compared against the highest age group of scores (i.e. 18y 00-18y 11m) (Martin, 2006). There are seven subtests of eighteen stimuli figures each, which assess seven key areas of visual perception. Each subscale consisting of eighteen figures including two example items and sixteen test items are arranged in order of increasing complexity (see App. A). The test is largely an untimed instrument with the exception of subtests for visual memory and visual sequential memory being allocated a five second presentation time per item. Response time is however not restricted for any of the items.

The Dynamic Occupational Therapy Cognitive Assessment instrument designed to assess the cognitive abilities and learning potential of children from ages 6 to 12 years via a dynamic mediation testing process. DOTCA-Ch, a criterion-referenced assessment, was designed to fill this need. Originally based on the Loewenstein Occupational Therapy Cognitive Assessment (LOTCA), an assessment for adults with neuropsychological deficits, the DOTCA-Ch represents an adapted and modified format that is appropriate for use with school-age children. The DOTCA-Ch battery consists of 22 subtests in 5 cognitive domains: Orientation, Spatial Perception, Praxis, Visuomotor Construction, and Thinking Operations. Construct validity was supported by comparing children with traumatic brain injury and learning disabilities to typically developing children, and ecological validity of children with attention deficit hyperactivity disorder by comparing performance on the DOTCA-Ch to the School Function Assessment. Results of the intraclass correlation coefficients analysis revealed very high reliability coefficients for all cognitive domains, ranging from .87 to .99.

The Behavior Rating Inventory of Executive Function (BRIEF) assesses problem behaviors associated with executive function. The form consists of 86 brief descriptions of behavior problems, the frequency of which teachers and parents are asked to rate as occurring either never, sometimes, or often. Responses are aggregated to form eight subscales (Inhibit, shift, emotional control, initiate, working memory, plan/organize, organization of materials and monitor scale). Examples of test items from each subscale are shown in the Appendix C and D. T-scores are calculated for each measure. The scales showed high internal consistency on the BRIEF (a=.80-.90) for both Teachers and Parents form. The moderate test-retest reliabilities for teachers BRIEF (.90-.92) and for the parent BRIEF (.80-.83). Interrater reliability of the teachers BRIEF is reported as .17-.28, and of the parents BRIEF as .32-.34. Both tools are reported to have evidenced for content of the items, convergence and divergence of their scores with other measures.

ELIGIBILITY:
Inclusion Criteria:

The participants have only dyslexia diagnosis, They aged between 7-12 years and They have a 90 and above IQ score (normal IQ).

Exclusion Criteria:

They have multiple conditions (neurological problems such as epilepsy) or primary psychiatric comorbidities (i.e. depression, anxiety, psychosis).

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2014-02-03 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
The Behavior Rating Inventory of Executive Function | This study pretest-posttest intervention and follow up (3 months) study was designed to assess the effects of the CBCT on children with dyslexia.
  The form consists of 86 brief descriptions of behavior problems, the frequency of which teachers and parents are asked to rate as occurring either never, sometimes, or often. Responses are aggregated to form eight subscales (Inhibit, shift, emotional control, initiate, working memory, plan/organize, organization of materials and monitor scale).
Test of Visual Perceptual Scale-3(TVPS-3); | This study pretest-posttest intervention and follow up (3 months) study was designed to assess the effects of the CBCT on children with dyslexia.
  The TVPS-3 was originally designed for children but the author Dr Gardner also reported statistically significant differences between three groups diagnosed as having either developmental delay, head injury or learning disability (Gardner, 1992). This test in its third edition has been revised by Martin for appropriate use in an adult population, with scores compared against the highest age group of scores (i.e. 18y00-18y11m)
The Dynamic Occupational Therapy Cognitive Assessment | This study pretest-posttest intervention and follow up (3 months) study was designed to assess the effects of the cognitive therapy on children with dyslexia.
  It instrument designed to assess the cognitive abilities and learning potential of children from ages 6 to 12 years via a dynamic mediation testing process. DOTCA-Ch, a criterion-referenced assessment, was designed to fill this need. Originally based on the Loewenstein Occupational Therapy Cognitive Assessment (LOTCA), an assessment for adults with neuropsychological deficits, the DOTCA-Ch represents an adapted and modified format that is appropriate for use with school-age children. The DOTCA-Ch battery consists of 22 subtests in 5 cognitive domains

SECONDARY OUTCOMES:
Executive Functions and Occupational Routines Scale (EFORTS) | This study pretest-posttest intervention and follow up (3 months) study was designed to assess the effects of the CBCT on children with dyslexia.
  The EFORTS, in the context of executive functions, was used to evaluate the performance levels in their child's daily routines. The EFORTS can be used to determine whether executive function deficit in children regardless of the diagnosis. The tool was developed as a parent's report about the executive control through their child's daily routines. Three subscales in this survey were defined as follows: 1) morning and evening routines; 2) play and leisure; and 3) social routines. Each item was rated with a Likert scale as follows: never (1), seldom (2), sometimes (3), frequently (4) and always (5). The encoding of the EFORTS helped with obtaining means for each of the functional routine and a final functional score (mean). The accrual score evaluation was calculated by the mean, giving a score for both total and subscales. Higher score, in each executive controlled daily routine activity have shown the better performance of the child.

IPD SHARING:
Plan to Share IPD: No
we have no plan to make individual participant data (IPD) available to other researchers.